CLINICAL TRIAL: NCT04397900
Title: A Blood Collection Study From Volunteers Who Have Recovered From COVID-19 Infection to Identify Immunogenic Viral Epitopes in SARS-CoV-2
Brief Title: Blood Collection Study From COVID-19 Convalescents Previously Hospitalized to Identify Immunogenic Viral Epitopes
Status: Completed | Type: Observational
Sponsor: TScan Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1586788
Record Dates: First submitted 2020-05-19; First posted 2020-05-21 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2020-05

CONDITIONS: Identify the Viral Epitopes of Memory CD8 T Cells From Individuals That Have Recovered From SARS-CoV-2 Infection; Determine Which SARS-CoV-2 Proteins Are Frequently Recognized by T Cells in Patients With Varying HLA Types

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The COVID-19 pandemic is a global emergency threatening to take millions of lives in the United States and around the world. There is no current vaccine strategy against COVID-19 infection caused by a novel coronavirus named SARS-CoV-2. Studies with a related coronavirus called SARS-CoV-1 that caused the SARS outbreak in 2003 indicated that memory CD8+ T cells recognizing viral epitopes persisted for more than 6 years post infection while neutralizing antibodies and memory B cells were short-lived and were undetectable after a short period of time (Tang et al., 2011; Peng et al., 2006; Channappanavar et al., 2014). Thus, including viral epitopes that are recognized by memory CD8+ T cells is imperative for vaccines that can provide long-term immunity against SARS-CoV-2. In this study, blood samples from COVID-19 patients who have recovered from the infection will be used to identify the viral epitopes recognized by their memory CD8+ T cells. This will be accomplished using a genome-wide, high-throughput screening technology developed at Harvard Medical School (Kula et al., 2019) and licensed by the study sponsor, TScan Therapeutics. A 24,000-member library that tiles across all ~100 viral isolates of SARS-CoV-2 that have been sequenced so far has already been synthesized at TScan. Blood samples from convalescent patients are urgently needed to identify T cell receptors and immunogenic viral epitopes on SARS-CoV-2. It is the hope that these data will inform development of a vaccine with the potential for long-lasting protection against SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory-confirmed diagnosis of COVID-19 performed by The Centers for Disease Control and Prevention (CDC) at a hospital using an FDA Emergency Use Authorized molecular assay for COVID-19
* Age =>18 years at time of diagnosis of COVID-19
* Time since discontinuation of isolation of =>14 day following CDC criteria
* Ability to understand and willingness to sign an informed consent document
* No anti-pyretic use for =>17 days
* Ability to undergo blood draw for 4 tubes of blood containing approximately 7.5 mL of blood each
* Ability to travel to an assigned lab for blood draw
* Ability to waive any claim to blood samples or data obtained for this study's purpose

Exclusion Criteria:

* Any serious medical or psychiatric disorder that would interfere with the subject's safety
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent
* Known blood disorder that would increase the risk of infection or bleeding from a simple phlebotomy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: COVID-19 convalescents previously hospitalized willing to donate blood. Both men and women and members of all races and ethnic groups are eligible for this protocol. It is expected that the mix of participants entering this study will reflect the demographics of the population affected by COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Identify the viral epitopes of memory CD8+ T cells from individuals that have recovered from SARS-CoV-2 infection. | JUL2020
Determine which SARS-CoV-2 proteins are frequently recognized by T cells in patients with varying HLA types. | JUL2020

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Atlantic Health System, Morristown, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang F, Quan Y, Xin ZT, Wrammert J, Ma MJ, Lv H, Wang TB, Yang H, Richardus JH, Liu W, Cao WC. Lack of peripheral memory B cell responses in recovered patients with severe acute respiratory syndrome: a six-year follow-up study. J Immunol. 2011 Jun 15;186(12):7264-8. doi: 10.4049/jimmunol.0903490. Epub 2011 May 16. PMID 21576510
- [Background] Peng H, Yang LT, Wang LY, Li J, Huang J, Lu ZQ, Koup RA, Bailer RT, Wu CY. Long-lived memory T lymphocyte responses against SARS coronavirus nucleocapsid protein in SARS-recovered patients. Virology. 2006 Aug 1;351(2):466-75. doi: 10.1016/j.virol.2006.03.036. Epub 2006 May 11. PMID 16690096
- [Background] Channappanavar R, Fett C, Zhao J, Meyerholz DK, Perlman S. Virus-specific memory CD8 T cells provide substantial protection from lethal severe acute respiratory syndrome coronavirus infection. J Virol. 2014 Oct;88(19):11034-44. doi: 10.1128/JVI.01505-14. Epub 2014 Jul 23. PMID 25056892
- [Background] Kula T, Dezfulian MH, Wang CI, Abdelfattah NS, Hartman ZC, Wucherpfennig KW, Lyerly HK, Elledge SJ. T-Scan: A Genome-wide Method for the Systematic Discovery of T Cell Epitopes. Cell. 2019 Aug 8;178(4):1016-1028.e13. doi: 10.1016/j.cell.2019.07.009. PMID 31398327
- [Background] Xu GJ, Kula T, Xu Q, Li MZ, Vernon SD, Ndung'u T, Ruxrungtham K, Sanchez J, Brander C, Chung RT, O'Connor KC, Walker B, Larman HB, Elledge SJ. Viral immunology. Comprehensive serological profiling of human populations using a synthetic human virome. Science. 2015 Jun 5;348(6239):aaa0698. doi: 10.1126/science.aaa0698. PMID 26045439